CLINICAL TRIAL: NCT05649579
Title: Efficacy and Safety of Dupilumab in Patients With Bullous Pemphigoid: a Multicenter Retrosepctive Study
Brief Title: Efficacy and Safety of Dupilumab in Patients With Bullous Pemphigoid
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Collaborators: Ruijin Hospital (Other); Chinese Academy of Medical Sciences (Other); West China Hospital (Other); Second Xiangya Hospital of Central South University (Other); Shandong Provincial Institute of Dermatology and Venereology (Other)
Responsible Party: Principal Investigator, Mingyue WANG, Principal Investigator, Peking University First Hospital
Other Study IDs: 2022Y446
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Bullous Pemphigoid
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Dupilumab — Duplimab was administered according to the guidelines of the atopic dermatitis treatment regimen, which involved the first dose of 600 mg followed by 300 mg every two weeks. Because of comorbidities or the side effects of corticosteroid, some patients used dupilumab in the initial course of treatment, while others added dupilumab when the traditional drugs proved ineffective. The discontinuation was a joint decision between treating dermatologists and patients. Concomitant medicine was decided by clinicians, depending on the assessing of disease status and patients' choices, and reduced according to international guidelines.
  Other Names: Dupixent

SUMMARY:
This study was designed to be a retrospective, multicentre, observational study to evaluate the efficacy and safety of dupilumab in the treatment of bullous pemphigoid and to find predictors of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Adult bullous pemphigoid patients treated with dupilumab between January 1, 2021, and July 31, 2022, at six leading dermatology departments in the Chinese Collaborative Network for Autoimmune Bullous Diseases.
* The diagnosis of BP requires clinical manifestations and immunological or pathological evidences.
* Dupilumab treatment should continue for at least 4 weeks and possibly longer.

Exclusion Criteria:

* Drug-induced BP, γ-1 pemphigoid
* Patients with less than 4 weeks of follow-up
* Patients were given any other biologicals within 6 months before the first dupilumab administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult bullous pemphigoid patients treated with dupilumab between January 1, 2021, and July 31, 2022, at six leading dermatology departments in the Chinese Collaborative Network for Autoimmune Bullous Diseases.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients reached disease control | within 4 weeks
  Disease control was defined as the point at which new lesions or pruritic symptoms cease to form and existing lesions start to heal.

SECONDARY OUTCOMES:
Complete remission rate | within 64 weeks
  Complete remission is defined as the absence of new or established lesions or pruritus while the patient is receiving minimal therapy or off therapy for at least 2 months.
Relapse rate | within 64 weeks
  Relapse was defined as the appearance of three or more new lesions a month or at least one eczematous lesion with a diameter >10cm or urticarial plaque that does not heal within one week, or the extension of established lesions or daily pruritus in a patient who has achieved disease control.
Adverse events | within 64 weeks
  Any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure.
Changes in BPDAI scores | from 0 to 64 weeks
  Disease severity was assessed using the bullous pemphigoid disease area index (BPDAI) score and was classified into mild (BPDAI≤19), moderate (20≤BPDAI≤56), and severe (BPDAI≥57).
Changes in itching NRS scores | from 0 to 64 weeks
  Pruritus was evaluated via itching numeric rating scale (NRS), ranging from 0 (no itch) to 10 points (worst imaginable itch).
Changes in serum anti-BP180 antibodies | from 0 to 64 weeks
Changes in serum anti-BP230 antibodies | from 0 to 64 weeks
Changes in serum total IgE | from 0 to 64 weeks
Changes in peripheral blood eosinophil count | from 0 to 64 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mingyue Wang, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China